CLINICAL TRIAL: NCT05455034
Title: Single-cell Sequencing of Bronchoalveolar Lavage Fluid to Guide the Treatment of Radiation Pneumonitis or Immune Checkpoint Inhibitor Pneumonitis
Brief Title: Single-cell Sequencing of BLF to Guide the Treatment of Radiation Pneumonitis or Immune Checkpoint Inhibitor Pneumonitis
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Xinqiao Hospital of Chongqing (Other)
Responsible Party: Principal Investigator, Jianguo Sun, Deputy director of oncology department, Clinical Professor, Xinqiao Hospital of Chongqing
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XQonc-019
Record Dates: First submitted 2022-06-30; First posted 2022-07-13 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Pneumonitis
Keywords: Single-cell Sequencing; Radiation Pneumonitis; Immune Checkpoint Inhibitor Pneumonitis; Bronchoalveolar Lavage Fluid
MeSH Terms: conditions — Pneumonia; Radiation Pneumonitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single-cell Sequencing of BLF to Guide the Treatment of Radiation Pneumonitis (Experimental): Single-cell Sequencing of BLF is detected before treatment, and then patients will receive the treatment of Radiation Pneumonitis according to the result.
  Interventions: Genetic: single-cell sequencing
- Single-cell Sequencing of BLF to Guide the Treatment of Immune Checkpoint Inhibitor Pneumonitis (Experimental): Single-cell Sequencing of BLF is detected before treatment, and then patients will receive the treatment of Immune Checkpoint Inhibitor Pneumonitis according to the result.
  Interventions: Genetic: single-cell sequencing

INTERVENTIONS:
Genetic: single-cell sequencing — Treatment is given according to the results of single-cell sequencing.

SUMMARY:
A multicenter, exploratory clinical research, to map the radiation or immune checkpoint inhibitor pneumonitis in patients with alveolar lavage single-celled map. Find out the pathogenesis and prevention strategies of radiation or immune checkpoint inhibitor pneumonitis. Specific treatment is given based on the recommendation of the treatment guidelines for radiation or immune checkpoint inhibitor pneumonitis and the results of single cell sequencing, which will become a new technology for clinical application.

DETAILED DESCRIPTION:
This study is a multicenter, exploratory clinical research, to map the radiation or immune checkpoint inhibitor pneumonitis in patients with alveolar lavage single-celled map. Find out the pathogenesis and prevention strategies of radiation or immune checkpoint inhibitor pneumonitis. Specific treatment is given based on the recommendation of the treatment guidelines for radiation or immune checkpoint inhibitor pneumonitis and the results of single cell sequencing, which will become a new technology for clinical application.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent has been signed, and according to the judgment of the investigator, the patient can comply with the study protocol and sign the written informed consent;
2. NSCLC patients who have been clinically diagnosed with RP or CIP after histopathologically confirmed radiotherapy or immunocheckpoint inhibitor treatment and have not received glucocorticoid or other drugs.
3. ≥18 years old, less than 75 years old;
4. ECOG PS score 0-3 in the Eastern Tumor Collaboration group;
5. Patients without contraindications to alveolar lavage;

Exclusion Criteria:

1. Poor patient compliance and violation of test regulations;
2. Liver and kidney dysfunction, such as myocardial infarction, angina pectoris, liver transaminase significantly increased;
3. Had any medical condition requiring systemic treatment with corticosteroids or other immunosuppressive drugs within 14 days prior to enrollment;
4. Severe infection occurred within 4 weeks prior to enrollment, including but not limited to hospitalization due to infection complications, bacteremia or severe pneumonia;
5. Severe chronic or active infections (including tuberculosis infection) requiring systemic (oral or intravenous) antibiotic treatment within 14 days prior to enrollment;
6. Untreated patients with chronic hepatitis B, HBV carriers with HBV DNA≥ 500 IU/mL, or patients with active hepatitis C virus (HCV) should be excluded. Note: Non-active hepatitis B, surface antigen (HBsAg) carriers, treated and stable hepatitis B carriers (HBV DNA & LT; 500 IU/mL), patients with cured hepatitis C could be enrolled;
7. Known history of HIV infection;
8. Received any other investigational drug or participated in any other clinical trial within 28 days.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Response rate | 8 weeks
  Tumor diameter is measured before and 8 weeks after treatment. Area alleviated by lung shadow or ground-glass changes more than 50% was significant; The alleviating area of lung shadow or ground-glass change was 20% ~ 50%. Area alleviated by shadow or ground-glass changes in lung after treatment. 20% or worse than before treatment is ineffective.

CONTACTS AND LOCATIONS:
Overall Officials: Jianguo Sun, doctor, Principal Investigator — Xinqiao Hospital
Locations (1):
- Xinqiao Hospital, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Papalexi E, Satija R. Single-cell RNA sequencing to explore immune cell heterogeneity. Nat Rev Immunol. 2018 Jan;18(1):35-45. doi: 10.1038/nri.2017.76. Epub 2017 Aug 7. PMID 28787399
- [Background] Liao M, Liu Y, Yuan J, Wen Y, Xu G, Zhao J, Cheng L, Li J, Wang X, Wang F, Liu L, Amit I, Zhang S, Zhang Z. Single-cell landscape of bronchoalveolar immune cells in patients with COVID-19. Nat Med. 2020 Jun;26(6):842-844. doi: 10.1038/s41591-020-0901-9. Epub 2020 May 12. PMID 32398875
- [Result] Grun D, van Oudenaarden A. Design and Analysis of Single-Cell Sequencing Experiments. Cell. 2015 Nov 5;163(4):799-810. doi: 10.1016/j.cell.2015.10.039. PMID 26544934